CLINICAL TRIAL: NCT00955344
Title: Increasing Primary Care Physician Colorectal Cancer Screening Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Carmen Guerra, M.D., Universirty of Pennsylvania School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K22CA133186-01 (NIH)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer screening; American Board of Internal Medicine Maintenance of Certification program; Currently enrolled in or plan to enroll in the American Board of Internal Medicine Maintenance of Certification program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based intervention (eToolbox) (Experimental): This arm will allow diplomats of the American Board of Internal Medicine to complete the Practice Improvement Module that will embed a link to the web-based intervention (eToolbox).
  Interventions: Behavioral: eToolbox
- Practice Improvement Module (Active Comparator): This arm will allow diplomats of the American Board of Internal Medicine to complete the Practice Improvement Module without any link to the Web-based eToolbox.
  Interventions: Behavioral: no link to eToolbox

INTERVENTIONS:
Behavioral: eToolbox — Participants randomized to the Web-based intervention will be automatically routed to a URL that will contain the Web-based intervention.
  Arms: Web-based intervention (eToolbox)
Behavioral: no link to eToolbox — Participants randomized to the Practice Improvement Module will not be automatically routed to a URL that will contain the Web-based intervention.
  Arms: Practice Improvement Module

SUMMARY:
The purpose of the study is to determine if a Web-based intervention increases physician rates of colorectal cancer recommendation rates in a group of physicians participating in the American Board of Internal Medicine's Maintenance of Certification Program. This study will also compare the content of practice improvement plans submitted by the diplomats in each study arm to determine the components of the plans that are associated with colorectal cancer rates.

DETAILED DESCRIPTION:
Colorectal cancer is the 2nd leading cause of cancer deaths in the U.S. Although colorectal cancer screening (CRCS) is effective, cost-effective and consistently recommended by clinical practice guidelines, only 57.3% of the adults over 50 years have been screened within the recommended interval. Preliminary research conducted by this PI demonstrates that approximately 90% of patients who have not had CRCS report that a doctors recommendation would motivate them to undergo screening. However, research also shows that physicians do not consistently recommend CRCS to each eligible patient. In this study the barriers of and facilitators to physician recommendation of CRCS are tested in the to proposed randomized controlled trial. The trial will pilot test an interactive, multifaceted, Web-based intervention (eToolbox) to increase primary care physician rates of CRCS. This application innovatively proposes to pilot test the eToolbox in the setting of the American Board of Internal Medicine (ABIM) Maintenance of Certification process within the Preventive Services Practice Improvement Module, a physician-directed measurement of their performance and quality improvement requirement for board re-certification.

ELIGIBILITY:
Inclusion Criteria:

* ABIM certification and have or plan to enroll in the Maintenance of Certification program
* Primary Care Physicians

Exclusion Criteria:

* Diplomats are not able to participate in this study if they are retired physicians, do not practice a primary care practice or who have already taken part in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening Rates | 3 years (2012)

SECONDARY OUTCOMES:
Content of practice improvement plan | 3 years (2012)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen E Guerra, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States